CLINICAL TRIAL: NCT03718182
Title: Can Vitamin D Supplementation in People With Crohn's Disease Improve Symptoms as an Adjunct Therapy? D-CODE Feasibility Randomised Controlled Trial
Brief Title: Can Vitamin D Supplementation in People With Crohn's Disease Improve Symptoms as an Adjunct Therapy?
Acronym: D-CODE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Birmingham (Other); Clinical Trials Research Centre (Unknown)
Responsible Party: Principal Investigator, Jane Fletcher, Nutrition Nurse Lead, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRK6542
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Crohn Disease; Vitamin D Deficiency
Keywords: vitamin D supplementation; quality of life; Inflammatory Bowel Disease Questionnaire IBDQ; Hepcidin
MeSH Terms: conditions — Crohn Disease; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: D-CODE is a two part trial entailing two vitamin D screening studies (winter and summer) and an interventional feasibility study.
  The vitamin D screening studies will take place during the winter and summer months to determine the prevalence of vitamin D deficiency in patients with CD throughout the seasons.
  In the intervention/feasibility stage D-CODE is an exploratory study for an open label, multi-site, superiority randomised controlled trial. Participants will be randomised to one of two parallel arms (A or B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - Cholecalciferol 400iu (Active Comparator): Vitamin D3 (Cholecalciferol) 400 iu. Daily oral capsule. To be taken for 24 weeks (6 months)
  Interventions: Dietary Supplement: Cholecalciferol
- Arm B - Cholecalciferol 3200iu/800iu (Experimental): Vitamin D3 (Cholecalciferol) supplement 3,200iu daily oral capsule. To be taken for 12 weeks (3 months).
  Then switch to vitamin D3 supplement 800iu daily oral capsule. To be taken for 12 weeks (3 months).
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — vitamin D3 daily oral supplement

SUMMARY:
There are around 115,000 people in the United Kingdom suffering with Crohn's Disease (CD). CD can cause inflammation and ulcers to develop anywhere within the gut. Symptoms of the disease include diarrhoea, abdominal pain and nutritional problems including vitamin D deficiency. Around half of people with CD are likely to have vitamin D deficiency. Research has shown that treating vitamin D deficiency in people with CD might help to improve the symptoms of the disease. However, there are no clear guidelines on how to detect or treat vitamin D deficiency in people with CD.

There will be two parts to the planned research involving three hospitals in Birmingham. Part 1 is a vitamin D screening study, where adults will be asked to have a finger-prick blood test to check their vitamin D levels. They will complete short diet and lifestyle questionnaires. Adults found to have vitamin D deficiency in part 1 may be invited to join part 2 of the research. Part 2 is a vitamin D supplementation study where participants will be given a daily vitamin D capsule to take by mouth for 6 months. They will be randomly allocated to 2 different groups with each group receiving a different dose of vitamin D. Participants will have blood tests at the start, after 3 months and after 6 months. They will complete quality of life questionnaires at the start and after 6 months. The last appointment will be a final follow up appointment after 9 months.

This research is important to help determine:

* Which dose of vitamin D is most effective at treating vitamin D deficiency in people with CD
* If symptoms of CD improve when vitamin D deficiency is treated.

ELIGIBILITY:
Inclusion Criteria:

1. VITAMIN D SCREENING STUDY

   Those:
   * With a confirmed diagnosis of Crohn's Disease (CD)
   * ≥ 18 years of age
   * Have provided written informed consent
2. VITAMIN D SUPPLEMENTATION FEASIBILITY TRIAL

Those:

* With a confirmed diagnosis of CD
* Identified as having Vitamin D deficiency < 50 nmol/L in the Winter screening study
* ≥ 18 years of age
* Already receiving treatment for CD as per National Institute for Health and Care Excellence (NICE) Guidance or those in remission and not currently receiving treatment but who continue to attend hospital out-patient appointments
* Have provided written informed consent

Exclusion Criteria:

1. VITAMIN D SCREENING STUDY

   * None
2. VITAMIN D SUPPLEMENTATION FEASIBILITY

Those:

* Currently receiving vitamin D, fish oil or multi-vitamin supplementation and unwilling to stop this to participate in the feasibility trial
* Currently receiving:

  * Bisphosphonates
  * Digitalis or other cardiac glycosides
  * Phenytoin
  * Barbituates (e.g. Amylobarbitone, Butobarbitone, Methyl Phenobarbitone, Pentobarbitone, Quinalbarbitone, Amylobarbitone)
  * Actinomycin
  * Imidazole
* With known hyperparathyroidism
* With known sarcoidosis
* With known renal disease or kidney stones
* With known hypercalcaemia (corrected serum calcium ≥2.60 mmol/L)
* With known underlying liver disease
* With known hypersensitivity to vitamin D supplements or any of the trial medication excipients
* Who are pregnant, breast feeding, trying to conceive or women of child-bearing age who decline to have a pregnancy test where applicable. Women who have had a hysterectomy, bilateral oophorectomy or early menopause will not require a pregnancy test.
* Individuals who have participated in a trial testing a medicinal product within 6 months preceding screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | 6 months
  Disease Related Quality of life patient reported outcome measure

SECONDARY OUTCOMES:
Euroquol EQ-5D-5L | 6 months
  Generic utility measure patient reported outcome

OTHER OUTCOMES:
Vitamin D 25(OH)D levels | 6 months
  Increase in serum vitamin D levels

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon C Cooper, Dr, Principal Investigator — Univeristy Hospital Birmingham NHS Trust
Locations (1):
- University Hospitals Birmingham NHS Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Fletcher J, Bedson E, Brown M, Hewison M, Swift A, Cooper SC. Protocol for an open-label feasibility study for a randomised controlled trial of vitamin D supplementation in Crohn's Disease patients with vitamin D deficiency: D-CODE Feasiblity study. Pilot Feasibility Stud. 2021 Mar 20;7(1):79. doi: 10.1186/s40814-021-00813-3. PMID 33743801